CLINICAL TRIAL: NCT05056922
Title: THRIVE-ASD: Telehealth Rapid Intervention for Externalizing Behaviors in ASD
Brief Title: Telehealth Rapid Intervention for Externalizing Behaviors in ASD
Acronym: THRIVE-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00114600; R41MC42775-01-00 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Disruptive Behavior; Externalizing Behavior; Parent-Child Interaction Therapy; Telehealth
MeSH Terms: conditions — Autism Spectrum Disorder; Problem Behavior | interventions — Therapeutics

STUDY DESIGN:
Masking Description: Research assistant coders will be blind to treatment condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-PCIT (Parent-Child Interaction Therapy) (Experimental)
  Interventions: Behavioral: Tele-PCIT
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Tele-PCIT — Families randomized to Tele-PCIT will receive a time-limited version of PCIT via telehealth. The first 5 sessions focus on the child directed interaction (CDI) phase. The first session includes a teaching session where the parent will learn PRIDE/"Do" skills and "Don't" skills. The next 4 CDI sessions include coaching where the therapist coaches the parent on the these skills within the context of play. The first PDI session includes a teaching session where parents will be given instructions for providing commands and timeout procedures. During the 4 PDI coaching sessions, the therapist coaches the parent through timeout procedures. Handouts are emailed to families throughout therapy. The treatment period is 12 weeks to complete the 10 sessions to account for scheduling challenges. Families will be provided a Bluetooth headset for sessions. Families who do not have access to a computer, tablet, or smartphone with internet access will be provided with a tablet for therapy use.
  Arms: Tele-PCIT (Parent-Child Interaction Therapy)
Behavioral: Treatment as Usual — Families randomized to Treatment-as-Usual (TAU) will receive brief feedback and psychoeducation during the baseline visit and will be provided with community resources and referrals as needed. The TAU procedures will reflect the level of care families receive after an ASD assessment or professional consultation in our own clinic. For addressing behavioral concerns specifically, families will be provided handouts on behavior management tips, given access to a webinar workshop reviewing basic behavioral parenting principles, and instructed to engage with available services. The Vanderbilt Treatment & Research Institute for ASD (TRIAD) Center offers a webinar series for managing challenging behaviors that parents will be directed to along with the Autism Speaks Challenging Behavior Toolkit handouts. The TAU period will be 12 weeks in length to match time specifications for the active treatment condition.
  Arms: Treatment as Usual

SUMMARY:
The purpose of this research study is to evaluate a time-limited version of Parent Child Interaction Therapy (PCIT) delivered via telehealth for young children with autism spectrum disorder (ASD) and disruptive behavior problems. Families will be randomly assigned to receive 10 sessions of Tele-PCIT or Treatment as Usual. Families will complete a baseline assessment, a post-treatment assessment, and a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 2:0 -6:11 years old
2. Have elevated levels of disruptive behavior problems as defined by the Eyberg Child Behavior Inventory
3. Have a diagnosis of ASD based on a positive Autism Diagnostic Observation Schedule (ADOS-2), a semi-structured parent interview, record review, and an ASD DSM-5 criteria checklist.
4. Have a receptive language age equivalent of at least 24 months as defined by the Peabody Picture Vocabulary Test
5. Are of low SES background defined by having primary Medicaid

Exclusion Criteria:

1. Presence of severe self-injurious behavior
2. Children who are receiving psychotropic medication and are not stable on their current medication regimen. Children receiving psychotropic medications who are on a stable regimen for one month will not be excluded.

Ages: 2 Years to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Child Behavior Problems as assessed by Eyberg Child Behavior Inventory (ECBI) | Pre-treatment to post-treatment (~12 weeks)
  The ECBI is a 36-item measure of disruptive behavior problems utilized across the PCIT literature. Parents will rate the frequency of child behaviors on a 7-point Likert scale. The ECBI yields a total raw score for intensity of behaviors and a normed T-score with higher scores indicating higher behavior problem severity. The cut-off for clinical significance is a raw score of 130.
Change in Child Behavior Problems as assessed by Eyberg Child Behavior Inventory (ECBI) | Pre-treatment to follow-up (~24 weeks)
  The ECBI is a 36-item measure of disruptive behavior problems utilized across the PCIT literature. Parents will rate the frequency of child behaviors on a 7-point Likert scale. The ECBI yields a total raw score for intensity of behaviors and a normed T-score with higher scores indicating higher behavior problem severity. The cut-off for clinical significance is a raw score of 130.
Change in Child Behavior Problems as assessed by Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) | Pre-treatment to post-treatment (~12 weeks)
  The SESBI is a 38-item measure of disruptive behavior utilized across the PCIT literature. Teachers will rate the current frequency of child behavior problems on a 7-point Likert scale and determine whether or not they find the behaviors to be problematic. The SESBI yields a total raw score for intensity of behaviors and a normed T-score with higher scores indicating higher behavior problem severity.
Change in Child Behavior Problems as assessed by Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) | Pre-treatment to follow-up (~24 weeks)
  The SESBI is a 38-item measure of disruptive behavior utilized across the PCIT literature. Teachers will rate the current frequency of child behavior problems on a 7-point Likert scale and determine whether or not they find the behaviors to be problematic. The SESBI yields a total raw score for intensity of behaviors and a normed T-score with higher scores indicating higher behavior problem severity.
Change in Child Compliance and Parent Interaction as assessed by Dyadic Parent-Child Interaction Coding System, 4th edition (DPICS-IV) | Pre-treatment to post-treatment (~12 weeks)
  The DPICS-IV observational paradigm and coding system is the gold standard for assessing parent and child observational outcomes across the PCIT literature. During each 5-minute parent-child situation (child-led, parent-led, clean-up), parents are provided standardized instructions via a bug-in-the-ear across a one-way mirror or video. All families are provided with the same set of standard toys during the observation. Each observation will be video recorded and subsequently coded for child compliance to commands and parenting "do" and "don't" skills by student research assistants who will be trained to research reliability and blinded to the child intervention status and timepoint.
Change in Child Compliance and Parent Interaction as assessed by Dyadic Parent-Child Interaction Coding System, 4th edition (DPICS-IV) | Pre-treatment to follow-up (~24 weeks)
  The DPICS-IV observational paradigm and coding system is the gold standard for assessing parent and child observational outcomes across the PCIT literature. During each 5-minute parent-child situation (child-led, parent-led, clean-up), parents are provided standardized instructions via a bug-in-the-ear across a one-way mirror or video. All families are provided with the same set of standard toys during the observation. Each observation will be video recorded and subsequently coded for child compliance to commands and parenting "do" and "don't" skills by student research assistants who will be trained to research reliability and blinded to the child intervention status and timepoint.
Change in Parenting Practices as assessed by Parenting Scale (PS) | Pre-treatment to post-treatment (~12 weeks)
  Parents will complete the PS, which has been consistently used across the PCIT literature as a measure of parenting practices. The PS is a 30-item measure, which yields a Total score representing an average of responses on all items, and individual scale scores for Laxness, Over-reactivity, and Negativity. A higher score on the scale scores and on the Total score indicates a greater level of reported problematic parenting discipline style.
Change in Parenting Practices as assessed by Parenting Scale (PS) | Pre-treatment to follow-up (~24 weeks)
  Parents will complete the PS, which has been consistently used across the PCIT literature as a measure of parenting practices. The PS is a 30-item measure, which yields a Total score representing an average of responses on all items, and individual scale scores for Laxness, Over-reactivity, and Negativity. A higher score on the scale scores and on the Total score indicates a greater level of reported problematic parenting discipline style.
Change in Parenting Stress as assessed by Parenting Stress Index-Short Form (PSI-SF) | Pre-treatment to post-treatment (~12 weeks)
  Parents will complete the PSI-SF, a 36-item measure yielding scores for a Total Stress scale. The PSI-SF is a widely used measure in ASD samples and has been used as an outcome measure in PCIT ASD studies. The PSI-SF yields a total raw score for stress level and a percentile score which describes parent stress relative to all parents assessed during the development and testing of the PSI. Scores above 80 are considered high stress scores.
Change in Parenting Stress as assessed by Parenting Stress Index-Short Form (PSI-SF) | Pre-treatment to follow-up (~24 weeks)
  Parents will complete the PSI-SF, a 36-item measure yielding scores for a Total Stress scale. The PSI-SF is a widely used measure in ASD samples and has been used as an outcome measure in PCIT ASD studies. The PSI-SF yields a total raw score for stress level and a percentile score which describes parent stress relative to all parents assessed during the development and testing of the PSI. Scores above 80 are considered high stress scores.
Change in Child Behavior Problems as assessed by Behavior Assessment System for Children-3rd Edition (BASC-3) | Pre-treatment to post-treatment (~12 weeks)
  Parents and teachers will complete the BASC-3, a broadband assessment that includes disruptive behavior domains including hyperactivity, aggression, and attention problems, in addition to a general externalizing behavior problems composite. The BASC-3 has excellent reliability and validity and has been utilized extensively across the ASD literature and in examinations of PCIT with ASD samples. The Preschool versions will be used for children 2 to 5 years old, and the Child version will be used for children 6:0+.
Change in Child Behavior Problems as assessed by Behavior Assessment System for Children-3rd Edition (BASC-3) | Pre-treatment to follow-up (~24 weeks)
  Parents and teachers will complete the BASC-3, a broadband assessment that includes disruptive behavior domains including hyperactivity, aggression, and attention problems, in addition to a general externalizing behavior problems composite. The BASC-3 has excellent reliability and validity and has been utilized extensively across the ASD literature and in examinations of PCIT with ASD samples. The Preschool versions will be used for children 2 to 5 years old, and the Child version will be used for children 6:0+.
Change in Child Behavior Problems as assessed by Disruptive Behavior Disorders Rating Scale (DBD) | Pre-treatment to post-treatment (~12 weeks)
  As a measure of disruptive behavior and symptoms of attention-deficit/hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD), parents and teachers will complete the DBD. The DBD contains 45items on a 4-point frequency scale. The DBD has been utilized in samples of preschoolers with ADHD and ODD, and in studies examining ADHD symptoms in samples of children with ASD.
Change in Child Behavior Problems as assessed by Disruptive Behavior Disorders Rating Scale (DBD) | Pre-treatment to follow-up (~24 weeks)
  The DBD is a 45-item measure of disruptive behavior and symptoms of attention-deficit/hyperactivity disorder (ADHD) and oppositional defiant disorder (ODD) that has been utilized in samples of preschoolers with ADHD and ODD, and in studies examining ADHD symptoms in samples of children with ASD. Parents and teachers will complete the DBD, rating each item on a four-point scale ranging from not at all (0) to very much (3).

SECONDARY OUTCOMES:
Parent Satisfaction with Tele-PCIT as assessed by Therapy Attitude Inventory (TAI) | Pre-treatment to post-treatment (~12 weeks)
  To assess treatment satisfaction, parents will complete the TAI, which is widely used in PCIT studies. Several questions will be added to the TAI to address parental satisfaction and openness regarding the telehealth delivery format for families in the Tele-PCIT condition. The TAI uses a Likert-type satisfaction scale and scores will be reported via descriptive statistics with 95% CIs within categories.
Impact of Barriers on Treatment Engagement as assessed by Barriers to Treatment Participation Scale (BTPS) | Pre-treatment to post-treatment (~12 weeks)
  Parents in Tele-PCIT will complete the BTPS at post-treatment to assess for the impact of barriers on treatment engagement throughout the intervention. The BTPS is a 44 item rating of how much parents agree with statements about their expectancies of barriers to treatment participation for their child, using a 5-point Likert scale (1=totally disagree, 5= totally agree). This measure has been used in other PCIT studies comparing engagement between clinic and telehealth delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT05056922/ICF_001.pdf